CLINICAL TRIAL: NCT04851821
Title: The Effectiveness of Phytotherapy in the Treatment of SARS-COV2 (COVID-19)
Brief Title: The Effectiveness of Phytotherapy in SARS-COV2(COVID-19)
Acronym: Quercetix
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, Professor, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Quercetix
Record Dates: First submitted 2021-02-06; First posted 2021-04-20 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: a Randomized Double-blind Study; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); PHYTOTHERAPIE
MeSH Terms: interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quercetix group (Experimental): Each patient included, after signing the consent, will have a treatment for ten days: one tablet twice a day 30 minutes before the meal.
  Interventions: Drug: Quercetin
- Placebo Group (Placebo Comparator): Each patient included, after signing the consent, will have a treatment for ten days: one tablet twice a day 30 minutes before the meal.
  Interventions: Drug: Quercetin

INTERVENTIONS:
Drug: Quercetin — Each patient included, after signing the consent, will have a treatment for ten days: one tablet times three per day 30 minutes before the meal.
  Other Names: PLACEBO

SUMMARY:
Quercetin is one of the flavonoids. Quercetin as well as rutin are recognized to be among the most active of the flavonoids. It is to quercetin that several medicinal plants, including ginkgo and St. John's Wort, owe part of their therapeutic effects. Often combined with vitamin C in supplements, it improves absorption by the body and delays its elimination.

Quercetin is extracted from a variety of plant sources, including the onion peel and seeds and pods of Dimorphandra mollis, a tree in the legume family native to South America.

At present, there is no scientific data to demonstrate the effectiveness of herbal medicine, regardless of the plant, to prevent or treat COVID-19. On the other hand, some plant-based food supplements have anti-inflammatory or immunomodulatory properties that may disrupt inflammatory defense mechanisms useful in fighting infections, and in particular against COVID-19.

DETAILED DESCRIPTION:
Type of study: a randomized, double-blind study using the Quercetine in the treatment of patients with SARS COV2 (covid-19) Quercetin is extracted from a variety of plant sources, including the onion peel and the seeds and pods of Dimorphandra mollis, a legume tree native to South America.

Although we are far from knowing everything about quercetin, its antioxidant, anti-inflammatory, and antihistamine (antiallergic) properties have been observed in numerous in vitro and animal studies.

History on quercetin In 1937, Albert Szent-Gyorgyi received a Nobel Prize for discovering vitamin C and flavonoids, as well as for exploring their biochemical properties. Originally, he gave the flavonoids the name "vitamin P" because of their effectiveness in reducing the permeability of blood vessels. This name was abandoned when it was realized that these substances were not really vitamins.

ELIGIBILITY:
Inclusion Criteria:

* all patients attending the emergency department for influenza-like illness.
* Being over 18 years old

Exclusion Criteria:

* Any patient requiring admission
* Non-consenting patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients | 10 DAYS
  Number of patients attending the emergency room

SECONDARY OUTCOMES:
disappearance of symptoms | 10 days
  Date of disappearance of symptoms present on admission
adverse reaction | 10 days
  Presence of an adverse reaction due to the administration of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia
Locations (1):
- Riadh Boukef, Sahloul, Sousse Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis Plan can be shared in supplimentary data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: In the publication of the article
Access Criteria: we will publish the Access criteria after the final Statistical analysis